CLINICAL TRIAL: NCT00902369
Title: A Study of AK106-001616 in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK106 II-01
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2010-07

CONDITIONS: Rheumatoid Arthritis
Keywords: AK106-001616
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AK106-001616

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AK106-001616 (Experimental)
  Interventions: Drug: AK106-001616
- Placebo (Placebo Comparator): Part1: AK106-001616 and Placebo
  Interventions: Drug: Placebo
- Active comparator (Active Comparator): Part2: AK106-001616 and Active comparator
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: AK106-001616 — Part1: Dose escalation Part2: Dose expansion
  Arms: AK106-001616
Drug: Placebo
  Arms: Placebo
Drug: Active comparator
  Arms: Active comparator

SUMMARY:
This will be a Phase II, multi-centre study consisting of 2 parts. Part 1: Clinical Pharmacology Study (drug-drug interaction between AK106-001616 and methotrexate) Part 2: Proof of Concept Study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA (class I to III)
* Stable dose of methotrexate (at least 12 weeks)

Exclusion Criteria:

* Pregnant or breastfeeding
* Abnormal screening laboratory test values considered to be clinically significant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Czechia (3):
  - Hlučín
  - Prague
  - Uherské Hradiště
- Germany (3):
  - Frankfurt am Main, Hesse
  - Berlin
  - Hamburg
- Hungary (2):
  - Budapest
  - Érd
- Vilnius, Lithuania
- Bucharest, Romania
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - Sheffield, South Yorkshire

REFERENCES:
- [Derived] Kozaki T, Tagashira M, Yamanishi K, Ellis B, Kayanoki T, Ooishi R, Sugiyama K, Matsuda S, Tsuruta K, Kohira T, Tsurui K. Evaluation of drug-drug interaction between the novel cPLA2 inhibitor AK106-001616 and methotrexate in rheumatoid arthritis patients. Xenobiotica. 2015;45(7):615-24. doi: 10.3109/00498254.2014.1000430. Epub 2015 Jan 12. PMID 25579091